CLINICAL TRIAL: NCT00576030
Title: Short-term Autonomic Effects of Caffeinated and Decaffeinated Espresso in Young Healthy Individuals
Brief Title: Action of Caffeinated and Decaffeinated Espresso on Autonomic Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof. Dr. H.-C. Deter, Dept of Psychosomatic Medicine and Psychotherapy, Benjamin Franklin Campus, Charité,Berlin
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: EA4/061/06; EA4/061/06
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2009-08

CONDITIONS: Influence of Espresso on Heart Rate Variability
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- H (Other): habitual coffee drinkers
  Interventions: Other: hab cof with water; Other: hab cof with dec espresso; Other: hab cof with caf espresso
- N (Other): non-habitual coffee drinkers
  Interventions: Other: non-hab cof with water; Other: non-hab cof with dec espresso; Other: non-hab cof with caf espresso

INTERVENTIONS:
Other: hab cof with water — habitual coffee drinker provided with water
  Arms: H
Other: hab cof with dec espresso — habitual coffee drinkers given decaffeinated espresso
  Arms: H
Other: hab cof with caf espresso — habitual coffee drinkers given caffeinated espresso
  Arms: H
Other: non-hab cof with water — non-habitual coffee drinkers given water
  Arms: N
Other: non-hab cof with dec espresso — non-habitual coffee drinkers given decaffeinated espresso
  Arms: N
Other: non-hab cof with caf espresso — non-habitual coffee drinkers given caffeinated espresso
  Arms: N

SUMMARY:
More than 80% of the population in the USA consume coffee each day. However there not many studies on change of heart rate variability and placebo effects after consumption of coffee.

In our study we aim to test the following hypotheses:

1. Habitual caffeinated espresso coffee drinkers show an increase in blood pressure, heart rate variability and parasympathetic activity (high frequency band) of the heart.
2. Non-habitual caffeinated espresso coffee drinkers show an increase of blood pressure. The heart rate variability and the parasympathetic activity of the heart will decrease.
3. Caffeinated or decaffeinated espresso induces comparable changes in habitual or non-habitual coffee drinkers.

ELIGIBILITY:
Inclusion Criteria:

* 18- 50 years old, healthy

Exclusion Criteria:

* Medication, obese(BMI > 30)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 70 minutes

SECONDARY OUTCOMES:
blood pressure | 70 min.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychosomatic Medicine and Psychotherapy, Charité University, Berlin, Germany